CLINICAL TRIAL: NCT05541874
Title: Establishment of 2D and 3D Primary Cell Cultures From Gastric and Gastroesophageal Junction Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and operative Intensive Care Medicine (CCM/CVK), Charité-Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: Gastric primary cell cultures
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Gastric and Gastroesophageal Junction Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators will establish primary cell cultures from surgically resected gastric and gastroesophageal junction cancer specimen that were collected between 06/2018 and 05/2021.

DETAILED DESCRIPTION:
Gastric cancer is among the leading causes of cancer-related death worldwide. Surgery or radiation monotherapy are applicable as treatment for localized tumors, however, the majority of patients are diagnosed in an advanced disease state requiring systemic therapy Chemotherapies are non-specific, affecting healthy tissues, and the overall response rate in gastric tumors is limited. As such, there is a large unmet medical need for targeted therapies against gastric tumors. Recent advances in the field of onco-immunology unraveled the mechanisms of immune response against cancer, leading to the development of immunotherapeutic strategies such as: immune check point inhibitors (ICIs), and advanced therapy medicinal products (ATMPs), e.g. chimeric antigen receptor (CAR) T cells. ICIs and CAR T cell therapy in particular have evolved as novel therapeutic cornerstones against hematological disease, but their efficacy against solid tumors remains poor. Accordingly, a minority of gastric cancer patients show durable responses to immunotherapies and there is currently no cellular immunotherapy available for gastric cancer. Further, gastric tumors are heterogeneous due to genomic changes, cellular composition, and the microenvironment, conferring a very variable response to immunotherapies. Thus, a personalized approach is needed, in order to understand individual resistance mechanisms and to predict which patients are most suitable for which therapy.

To address this need, test systems resembling patient-specific tumor biology are required. Cell lines lack 3D context and lose their genetic fidelity through passaging. Patient-derived murine xenograft models provide 3D environment and multi-organ context, but the xeno-environment hampers reliability and translatability. The investigators envision patient-derived tumor organoids as a superior model, as they are 3D self-organizing structures which reflect the tumor complexity. In addition, they have the potential to serve as patient avatars and preclinical models to predict the efficacy of therapies.

In this study, the investigators will establish patient-derived organoids and to study individual tumor biology and as testing platforms for (immune-) therapies. The investigators further investigate the individual biology of the patients tumors and healthy tissues to not only understand the heterogeneous mechanisms of gastric cancer but also the heterogeneous mechanisms of healthy gastric tissue in the fields of infectiology and immunology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric or gastroesophageal junction cancer

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric or gastroesophageal junction cancer
Sampling Method: Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Establishing primary cell cultures from gastric and gastroesophageal junction cancer. | 06/2018-05/2021
  With this study, want to establish an efficient protocol for the generation of primary cell cultures from gastric and gastroesophageal junction cancer.
  Primary outcome is the success rate of primary cell culture establishment.

SECONDARY OUTCOMES:
Investigating mechanisms of disease in the individual patient. | 06/2018-05/2021
  With this study, we want to generate primary cell cultures that represent the patients individual tumor. We want to use the primary cell cultures to model individual resistance mechanisms to therapies, immunotherapies like CAR T cells in particular.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof, Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No